CLINICAL TRIAL: NCT00619905
Title: A Randomized, Double-Blind, Placebo-Controlled, Cohort Dose Escalation Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ACZ885 (Anti-Interleukin-1Beta Monoclonal Antibody) in Patients With Active Rheumatoid Arthritis (RA) Despite Ongoing Treatment With Methotrexate (MTX) 15 mg or More Weekly for at Least 3 Months.
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ACZ885 in Patients With Rheumatoid Arthritis With Ongoing Treatment With Methotrexate
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CACZ885A2101
Record Dates: First submitted 2008-02-08; First posted 2008-02-21 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2008-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Anti-interleukin-1 beta; ACZ885
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ACZ885
- 2 (Placebo Comparator)
  Interventions: Drug: ACZ885

INTERVENTIONS:
Drug: ACZ885
  Arms: 1
Drug: ACZ885
  Arms: 2

SUMMARY:
This study assessed the long-term safety and tolerability of ACZ885 in patients with rheumatoid arthritis, as well as long-term efficacy, long-term preservation and/or improvement of joint structure and bone mineral density, and long term maintenance of health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18.5 - 65/75 years (depending on the dose group).
* Diagnosis of rheumatoid arthritis (ACR 1987 revised classification for criteria for RA) with a disease duration of at least 6 months prior to randomization.
* Active disease at screening and baseline evaluation (same evaluator) ) with more than 6 tender and 6 swollen joints of 28 examined (including any effused joint) and either a) Westergren erythrocyte sedimentation (ESR) ≥ 28 mm/hour, or b) CRP ≥ 6 mg/L.
* Patients should have failed at least 1 DMARD in the past, but should not be deemed "refractory to all therapies"
* Patients should have a current treatment regimen of ≥ 15 mg methotrexate/week and with the current dose stable for approximately 3 months.
* Patients were required to have an otherwise stable RA therapeutic regimen, consisting of either a stable dose of NSAIDs and/or a stable dose of oral corticosteroids (prednisone or equivalent < 10 mg daily) for at least 4 weeks prior to randomization.

Exclusion Criteria:

* Previous treatment with anti-TNF-α antibody therapy (or other biological therapy) within appropriate timeframe (considering the half life of the compound)
* Patients who have received intra-articular or systemic corticosteroid injections having been required for treatment of acute RA flare (not being part of a regular therapeutic regimen) within four weeks prior to randomization OR require narcotic analgesics other than those accepted by the investigator for analgesia (e.g., codeine, tramadol, dextropropoxyphene)

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2003-12; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Adverse events and infections occurrence throughout the study. | throughout the study
Presence of anti-ACZ885 antibodies in serum at baseline, Days 43, 71 and end of study (Day 113). | throughout the study

SECONDARY OUTCOMES:
ACR response criteria [including joint counts, patient/investigator disease activity and pain assessment, acute phase reactants (ESR and CRP) and a Health Assessment Questionnaire (HAQ)] . | throughout the study
Disease Activity Score (DAS) at baseline and Days 43 and 113. | throughout the study
Quantification of IL-1B, IL-6, and C-reactive protein (CRP), matrix metalloproteinases (MMPs) 1 and 3, and c-telopeptide of Type I collagen (Crosslaps), at Week 7 versus baseline. | throughout the study
Serum concentrations of ACZ885 at each visit. | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis investigator site
Locations (10):
- Germany (6):
  - Novartis Investigator Site, Berlin
  - Novartis Investigator Site, Cologne
  - Novartis Investigator Site, Hamburg
  - Novartis Investigator Site, Leipzig
  - Novartis Investigator Site, Munich
  - Novartis Investigator Site, Ratingen
- Netherlands (2):
  - Novartis Investigator Site, Leiden
  - Novartis Investigator Site, Nijmegen
- Switzerland (2):
  - Novartis Investigator Site, Bern
  - Novartis Investigator Site, Geneva

REFERENCES:
- [Derived] Alten R, Gram H, Joosten LA, van den Berg WB, Sieper J, Wassenberg S, Burmester G, van Riel P, Diaz-Lorente M, Bruin GJ, Woodworth TG, Rordorf C, Batard Y, Wright AM, Jung T. The human anti-IL-1 beta monoclonal antibody ACZ885 is effective in joint inflammation models in mice and in a proof-of-concept study in patients with rheumatoid arthritis. Arthritis Res Ther. 2008;10(3):R67. doi: 10.1186/ar2438. Epub 2008 Jun 5. PMID 18534016